CLINICAL TRIAL: NCT02423382
Title: Measurement of the Retinal Oxygen Saturaiton After Long-term Silicon Oil Tamponade With Oxymap
Brief Title: Measurement of the Retinal Oxygen Saturaiton After Long-term Silicon Oil Tamponade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Bingsheng Lou, DR., Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLT201405
Record Dates: First submitted 2015-04-14; First posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Retinal Detachment
Keywords: silicone oil; retinal saturation; retinal blood flow; retinal detachment
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3-6 months group (Other): In this group, the patients will recieve the surgery of silicone oil removal when silicone oil has been filled into eye for 3-6 months.
  Interventions: Procedure: Silicone oil removal
- 6-9 months (Other): In this group, the patients will recieve the surgery of silicone oil removal when silicone oil has been filled into eye for 6-9 months.
  Interventions: Procedure: Silicone oil removal
- >9 months (Other): In this group, the patients will recieve the surgery of silicone oil removal when silicone oil has been filled into eye for more than 9 months.
  Interventions: Procedure: Silicone oil removal

INTERVENTIONS:
Procedure: Silicone oil removal — The patients in each group will receive the same procedure of silicone oil removal.

SUMMARY:
The purpose of this study is to evaluate the effects of long-term tamponade with silicone oil on retinal saturation with Oxymap.

DETAILED DESCRIPTION:
Silicone oil is the first choice treatment for long-term vitreous replacement in complicated cases of retinal detachment. However, it will cause various problems for permanent tamponade, such as keratopathy, glaucoma, cataracts, and silicone oil emulsification3. In addition, silicone oil has the potential to cause retinal toxicity. Moreover, the gravity and mechanical pressure of the silicone oil on the retina may influence retinal blood flow and, and the presence of silicone oil in the vitreous cavity may block the oxygen exchange between the retinal surface and the vitreous humor, resulting in the metabolic disturbance of the retina. In this study, the investigators utilized a noninvasive measurement (Oxymap, Reykjavik, Iceland) to evaluate the effect of silicone oil tamponade on oxygen saturation and diameter in retinal vessels in complicated retinal detachment cases.

ELIGIBILITY:
Inclusion Criteria:

* initial silicone oil tamponade duration of more than 3 months
* transparent reflecting media
* intraocular pressure (IOP) between 11 and 21mmHg
* complete retinal re-attachment
* healthy contralateral eye.

Exclusion Criteria:

* severe refractive media opacity (serious keratoleukoma and cataracts)
* silicone oil emulsification
* ocular hypertension
* retinal detachment
* retinal scar within the main vascular arch
* any ocular disease and any history of surgery in the contralateral eye
* any type of systemic disease
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2014-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The changes from baseline in the retinal oxygen saturation by Oxymap at 2 months | 1 day before silicone oil removal and 2 months after silicone oil removal.

SECONDARY OUTCOMES:
The changes from baseline in the retinal vessel width by Oxymap at 2 months | 1 day before silicone oil removal and 2 months after silicone oil removal.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Lin, MD, Ph.D, Study Chair — Zhongshan Ophthalmic Center at Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China